CLINICAL TRIAL: NCT03390543
Title: The Effect of Simple Needle Guide Device for Ultrasound-guided Internal Jugular Vein Catheterization in Cardiac Surgical Patients: a Randomized-controlled Trial
Brief Title: The Effect of Simple Needle Guide Device for Ultrasound-guided Internal Jugular Vein Catheterization in Cardiac Surgical Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study plan is cancelled because of difficulties in the progress of the study.
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 1-2017-0047
Record Dates: First submitted 2017-12-20; First posted 2018-01-04 (Actual); Last update posted 2019-01-17 (Actual); Status verified 2019-01

CONDITIONS: Cardiac Surgery

STUDY DESIGN:
Intervention Model Description: 1. sono with simple needle guide device group
  2. sono only group
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: participants, investicator, outcome assessors will be blinded for group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Device group (Group D) (Experimental): Arm Description: Patients in this group are assigned to receive internal jugular vein catheterization guided by ultrasound and simple needle guide device.
  Interventions: Device: Sono with Device
- sono only group (Group S) (Placebo Comparator): Patients in this group are assigned to receive internal jugular vein catheterization guided by ultrasound without simple needle guide device.
  Interventions: Device: sono only

INTERVENTIONS:
Device: Sono with Device — In Group D, simple needle guide device was attached to the sono probe. Device was designed to assist the detection of the puncture site. After induction of anesthesia, both the device and sono-guided internal jugular vein catheterization was performed.
  Arms: Device group (Group D)
Device: sono only — In Group S, simple needle guide device was not attached to the sono probe. After induction of anesthesia, only sono-guided internal jugular vein catheterization was performed.
  Arms: sono only group (Group S)

SUMMARY:
The purpose of this study is to evaluate the effect of simple needle guide device for ultrasound-guided internal jugular vein catheterization in cardiac surgical patients

ELIGIBILITY:
Inclusion Criteria:

1. adult ( ≧19 years old)
2. patients undergoing elective cardiac surgery

Exclusion Criteria:

1. emergency surgery
2. patients under cervical immobilization
3. anatomical abnormality
4. infection or hematoma at puncture site
5. patients who did not need internal jugular vein catheterization

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-01-17 (Estimated); Primary Completion 2018-11-30 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
First access success rate | up to 5 minutes after insertion of puncture needle
  First access success rate was defined as the number of sono-guided catheterization obtained within first attempt.

SECONDARY OUTCOMES:
insertion time | 10 minutes after the beginning of the procedure
  defined as the time in seconds between the beginning of the procedure and guide-wire insertion
complication rate | 24 hours after surgery
  incidence of Pneumothorax, Haemothorax, Hydrothorax, carotid artery puncture, Hematoma, Malpositions, puncture of posterior wall of internal jugular vein
ease of procedure | 10 minutes after the beginning of the procedure
  In order to measure the degree of difficulty felt by the subjects during the procedure, a 100mm visual analogue scale was used to measure 10 difficulty levels (100mm; ease, 0mm ; difficult)
The number of attempts | 10 minutes after the beginning of the procedure
  The number of attempts was counted each time a subject inserted a guide needle into the neck surface, followed by withdrawal, redirection, or reinsertion.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Yonsei University College of Medicine, Seoul, Korea, South Korea

IPD SHARING:
Plan to Share IPD: No